CLINICAL TRIAL: NCT05585216
Title: The Efficacy of PRP Combined With Leg Swing and Quadriceps Strengthening Exercise to Treat Knee Osteoarthritis
Brief Title: The Efficacy of PRP Combined With Exercise to Treat Knee Osteoarthritisq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QIE001
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Platelet-rich Plasma; Physical Exercise; Knee Osteoarthritis
MeSH Terms: conditions — Motor Activity; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP combined with leg swing and quadriceps strengthening exercise (Experimental): Group A received twice intra-articular injection of platelet-rich plasma (2 ml, 2 weeks apart) and regular leg swing and quadriceps strengthening exercise for three months.
  Interventions: Drug: platelet-rich plasma
- intra-articular combination injections of PRP and HA (Active Comparator): Group B received twice intra-articular combination injections of PRP (2 ml) and HA (2 ml) every 2 weeks.
  Interventions: Drug: platelet-rich plasma

INTERVENTIONS:
Drug: platelet-rich plasma — intra-articular combination injections of platelet-rich plasma and hyaluronic acid or intra-articular combination injections of PRP combined with leg swing and quadriceps strengthening exercise

SUMMARY:
Objective. In this study, the investigators aimed to investigate the efficacy of combined a single platelet-rich plasma (PRP) and physical exercise (leg swing and quadriceps strengthening exercise) versus PRP and hyaluronic acid (HA) combination therapy. Methods. One hundred and six patients with grade Ⅱ-Ⅲ Knee osteoarthritis (KOA) according to the Kellgren-Lawrence classification were randomly divided into intra-articular injection of PRP combined with leg swing and quadriceps strengthening exercise (group A) and intra-articular combination injections of PRP and HA (group B). Patients in group A received twice intra-articular injection of PRP (2 ml, 2 weeks apart) and regular leg swing and quadriceps strengthening exercise for 3 months. Patients in group B received twice intra-articular combination injections of PRP (2 ml) and HA (2 ml) every 2 weeks. The primary outcome measures were Visual Analogue Scale (VAS) and Western Ontario and McMaster Universities (WOMAC) score. The second outcomes included single leg stance test (SLS) and functional activity by 2 minutes walking test (2MWT) and time up and go test (TUGT). All outcomes were evaluated at baseline and after 1,3,6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 45 years old;
* KOA was diagnosed according to the American College of Rheumatology Classification Criteria;
* patients with the Kellgren-Lawrence grade (K-L grade) for KOA of Ⅰ-Ⅲ;
* a history of symptoms more than three month, and patients with independent mobility.

Exclusion Criteria:

* lower limb axial deviation large than 5° (valgus and varus knee);
* patients with diabetes mellitus, sever cardiovascular disease, immunosuppressive status, mental illness or other diseases than might affect the results;
* injections or other invasive treatments into the lower extremities were used in the past three months;
* patients willing to follow the doctor's recommendation for exercise training;
* patients with previous knee fracture or malignancy;
* patients with a previous history of hip or knee joint surgery;
* patients participating in hip or knee muscle strengthening in the past 3 months;
* patients did not complete the intervention strategies or regular follow-up.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 12 months
  Degree of knee pain during treatment
Western Ontario and McMaster Universities (WOMAC) score | 12 months
  Severity of knee osteoarthritis

SECONDARY OUTCOMES:
single leg stance test (SLS) | 12 months
  Assess the patient's balance
2 minutes walking test (2MWT) | 12 months
  Assess the patient's functional activity
time up and go test (TUGT) | 12 months
  time up and go test (TUGT)

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No